CLINICAL TRIAL: NCT01362699
Title: A Single Center, Randomized, Double Blind, Placebo Controlled, Parallel Group Study of the Efficacy of JNJ 31001074 on Cue Induced Craving for Alcohol in Adult Subjects With Alcohol DependenceH3 Alcoholism
Brief Title: Effect of JNJ 31001074 on Urge to Drink in Alcohol-Dependent Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Re-prioritization lead to study cancellation.
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Compound Development Team Leader, Janssen Research & Development, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018802; 31001074ALC2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-05-19; First posted 2011-05-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Alcoholism
Keywords: Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders; Alcohol Dependence; JNJ-31001074; Bavisant
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders | interventions — bavisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-31001074 (Experimental)
  Interventions: Drug: JNJ-31001074
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-31001074 — Type=exact number, unit=mg, number=3, form=tablet, route=oral use. One tablet once daily for 7 days.
  Arms: JNJ-31001074
Drug: Placebo — Form=tablet, route=oral administration. One tablet once daily for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether JNJ-31001074 taken for 7 days reduces the urge to drink alcohol in alcohol-dependent study participants who are not seeking treatment.

DETAILED DESCRIPTION:
This study will evaluate whether JNJ 31001074 reduces the urge to drink alcohol in non treatment seeking, adult study participants with current alcohol dependence. Individuals who meet criteria for study participation will be randomly assigned to one of two treatment groups (tablets containing JNJ 31001074 or placebo tablets with no active ingredients) in a 1:1 ratio. Treatment group assignment will not be known by study participants or study staff. Baseline assessments will be recorded and participants will return to the clinic for testing on the last day of taking their assigned study medication for 7 days at home. Alcohol use is not allowed for 3 days prior to this end-of-dosing testing. During this test, their urge to drink alcohol and their mood will be measured while they view various computer images and then are presented with (but do not drink) either a favorite alcoholic beverage or water. Other measures will be collected during the study to evaluate the safety and tolerability of the study medication, including potential effects on sleep, as well as measures of thinking and cigarette smoking. Participants will return for a follow-up visit approximately 1 week after finishing the study medication and completing the clinic assessment above. Study participants will take one 3-mg tablet of JNJ-31001074 or matching placebo in the morning, preferably with food, for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Currently alcohol dependent but not seeking treatment
* Meets study criteria for amount of alcohol consumed
* Otherwise healthy
* Urge to drink increased by the presence of alcohol
* Able to complete and understand questionnaires and study procedures in English
* Willing and able to comply with the study requirements, including a 3-day period of alcohol abstinence and use of highly effective contraceptive methods
* Signed informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding
* Significant medical or psychiatric conditions other than alcohol dependence
* History of, or at risk of, medically significant alcohol withdrawal syndrome
* Dependent on substances other than alcohol , nicotine or caffeine
* Smokes more than 1 pack of cigarettes per day or consumes more than 500 mg caffeine per day
* Has glaucoma, cataracts, a history of eye inflammation, eye injury, or eye surgery other than to correct vision
* Treatment in the past 1 month prior to screening with disulfiram (Antabuse), acamprosate (Campral), naltrexone (ReVia or Vivitrol), or topiramate (Topamax)
* In need of or currently taking any psychoactive medications

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Urge to drink | 1 week

SECONDARY OUTCOMES:
The number of patients reporting adverse events as a measure of safety and tolerability | Up to approximately 15 days
Abnormal findings from eye exams performed as a measure of safety and tolerability | Up to approximately 8-15 days
Vital signs measurements as a measure of safety and tolerability | Up to approximately 15 days
Electrocardiograms as a measure of safety and tolerability | Up to approximately 15 days
Clinical Laboratory tests as a measure of safety and tolerability | Up to approximately 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- La Jolla, California, United States